CLINICAL TRIAL: NCT00333203
Title: Clinical Evaluation of the Safety of Next Generation Ophthalmic Irrigating Solution Compared to BSS Plus for Use During Surgery for Removal of Epimacular Membrane and Vitrectomy
Brief Title: Next Generation Ophthalmic Irrigating Solution Posterior Segment Study
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: C-04-18
Record Dates: First submitted 2006-06-01; First posted 2006-06-02 (Estimated); Last update posted 2012-03-05 (Estimated); Status verified 2012-03

CONDITIONS: Eye Diseases
Keywords: epimacular membrane
MeSH Terms: conditions — Eye Diseases; Epiretinal Membrane | interventions — glutathione-bicarbonate-Ringer solution

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- NGOIS (Experimental)
  Interventions: Drug: Next Generation Ophthalmic Irrigating Solution (NGOIS)
- BSS Plus (Active Comparator)
  Interventions: Other: BSS Plus

INTERVENTIONS:
Drug: Next Generation Ophthalmic Irrigating Solution (NGOIS) — Volume sufficient to irrigate adequately during cataract surgery
  Arms: NGOIS
Other: BSS Plus — Volume sufficient to irrigate adequately during cataract surgery
  Arms: BSS Plus

SUMMARY:
The purpose of this study is to evaluate the safety of Next Generation Ophthalmic Irrigating Solution (NGOIS) compared to BSS PLUS for use during surgery for removal of epimacular membrane and vitrectomy.

ELIGIBILITY:
Inclusion Criteria:

* Patients of any race and sex, with an epimacular membrane who would benefit from vitrectomy and membrane removal.
* Other protocol-defined inclusion criteria may apply.

Exclusion Criteria:

* Under 18 years of age.
* Other protocol-defined exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 369 (Actual)
Dates: Start 2005-10; Primary Completion 2006-03 (Actual); Study Completion 2006-03 (Actual)

PRIMARY OUTCOMES:
Best-corrected logMAR visual acuity

SECONDARY OUTCOMES:
Intraocular pressure (IOP)

CONTACTS AND LOCATIONS:
Locations (1):
- United States, Fort Worth, Texas, United States